CLINICAL TRIAL: NCT05338983
Title: Effect of Different Approaches of Delivering Local Dental Anesthesia on Pain Perception in Children. A Double Blinded Randomized Controlled Clinical Trial.
Brief Title: Effect of Different Approaches of Delivering Local Dental Anesthesia on Pain Perception in Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Dental local anesthesia pain
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Pain; Local Anesthetics; Epinephrine; Vibration
MeSH Terms: conditions — Pain | interventions — Anesthetics, Local; Sodium Bicarbonate; Mepivacaine

STUDY DESIGN:
Intervention Model Description: Children will be divided into 4 equal groups, 20 children each. Three experimental groups, and a(control group) . The 4 groups will be randomly allocated for each technique using block technique of simple random sampling. Randomized block designs are constructed to reduce noise or variance in the data.
  Every block will include the equal number of the four groups (three experimental and one control).
Who Masked: Participant, Investigator
Masking Description: The observer and the recipients will be blinded to the study group to avoid bias (double blind randomized controlled trial)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control: Traditional local anesthesia (Active Comparator): After proper isolation and drying of the injection site, the topical anesthetic gel (20% benzocaine) will be applied to the injection site using sterile cotton tipped applicator for 60 seconds, then the anesthesia (2% mepivacaine hcl with 1:100000 epinephrine) will be administere
  Interventions: Drug: Topical anesthetic; Drug: Mepivacaine Hydrochloride
- Group A (Warm group) (Experimental): The topical anesthetic gel (20% benzocaine) will be applied to the injection site using sterile cotton tipped applicator for 60 seconds. The cartridge of anesthetic solution will be placed in the baby bottle warmer in 300 ml of cold water (21°C). The anesthetic fluid will be warmed to reach 37°C (98.6°F) ,then the local anesthesia((2% mepivacaine hcl with 1:100000 epinephrine) will be administered
  Interventions: Drug: Topical anesthetic; Device: Avent baby bottle warmer; Drug: Mepivacaine Hydrochloride
- Group B (Buffered group) (Experimental): The topical anesthetic gel (20% benzocaine) will be applied to the injection site for 60 seconds,0.1ml of 8.4% of sodium bicarbonate will be removed from the 50 ml vial by one ml insulin syringe and directly injected into the local anesthetic cartridge. The cartridge will be shacked 5 times to mix the solution, then the local anesthesia(2% mepivacaine hcl with 1:100000 epinephrine) will be administered.
  Interventions: Drug: Topical anesthetic; Drug: Sodium bicarbonate; Drug: Mepivacaine Hydrochloride
- Group C (Buzzy group) (Experimental): After the child setting on the dental chair,(20% benzocaine) topical anesthetic gel will be applied to the injection site for 60 seconds. He will be familiar with the Buzzy device by explaining how it works in simple words. The wings of the device will be kept in the freezer. Once the child is ready, the frozen wings will be attached to the device and Buzzy will be placed extra-orally above the area/cheek where local anesthetic will be delivered. Once Buzzy is being held in place by hand, press the button or switch on the top of Buzzy, then the anesthesia (2% mepivacaine hcl with 1:100000 epinephrine) will be administered.
  Interventions: Drug: Topical anesthetic; Device: Buzzy device; Drug: Mepivacaine Hydrochloride

INTERVENTIONS:
Drug: Topical anesthetic — 20% Benzocaine gel will be applied on the area of infiltration
Device: Avent baby bottle warmer — Warming device
  Arms: Group A (Warm group)
Drug: Sodium bicarbonate — 0.1ml of 8.4% of sodium bicarbonate will be removed from the 50ml vial by one ml insulin syringe , directly injected into the local anesthetic cartridge and will be shacked 5 times to mix the solution.
  Arms: Group B (Buffered group)
Device: Buzzy device — Bee-shaped apparatus consisting of two parts: the main vibrating body of a bee and detachable ice wings.
  External application of Buzzy device during administration of dental anesthetic.
  Arms: Group C (Buzzy group)
Drug: Mepivacaine Hydrochloride — Mepivacaine HCL 2% with Epinephrine 1:100,000 Local Anesthetic. Local Dental anesthetic infiltration

SUMMARY:
The aim of the study is to compare the efficacy of three different approaches of local anesthesia (LA) administration (Warm[37°C] LA, Buffered LA, and BUZZY device) on pain perception to young children ( 6-12 years old) using sound -eye -motor and Wong-Baker FPR scales.

DETAILED DESCRIPTION:
Pain is an unpleasant sensory and emotional experience associated with actual or potential tissue damage.In pediatric dentistry, the injection of local anesthesia is the most common cause of fear and expected to be painful.So, an effective pain control significantly contributes to an optimal dental treatment in pediatric dentistry.Proper pain prevention may enhance the child's cooperation by building dentist-child trust and reducing fear and/or anxiety during the current or future visit(s). The purpose of this study is to compare the efficacy of three different approaches of LA administration(Warm[37°C] LA, Buffered LA, and BUZZY device) on pain perception to young children ( 6-12 years old) using sound -eye -motor and Wong-Baker FPR scales. This study will be conducted on 80 children aged between 6-12 years from pediatric dental clinic, Faculty of Dentistry, Mansoura University. Children will be divided to 4 equal groups, 20 children each. Three experimental groups, and a (control group) . The 4 groups will be randomly allocated for each technique using block technique of simple random sampling .Randomized block designs are constructed to reduce noise or variance in the data.

Every block will include the equal number of the four groups (three experimental and one control).

ELIGIBILITY:
Inclusion Criteria:

1. Children requiring maxillary infiltration LA for dental treatment.
2. Cooperative children (positive or definitely positive on Frankel's scale).
3. Children are in apparently good health and not taking any medications that will alter their pain perception.
4. Children have no history of allergy to Mepivacaine

Exclusion Criteria:

1. The person responsible does not authorize the participation of the child as a research volunteer.
2. Be using pain modulating drugs.
3. Patients with a history of hypersensitivity to local anesthetics.
4. Patients with a history of systemic diseases.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Behavoir | During the anesthetic procedure
  The pain will be analyzed by sound ,eye motor scale An assistant will be trained to measure and calibrate the SEM scale. The assistant will be blinded to the study group to avoid bias.
Self-perception of pain | Immediately after anesthesia
  The pain will be analyzed by the Wong Baker Faces scales
  . A set of six cartoon faces will be shown to the child with varying facial expressions ranging from a very smiling face to a very sad face. A brief explanation will be given to the child about each face after which the child will be instructed to choose the face that will describe his/ her feelings while receiving local anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Sahar H Zidan, Principal Investigator — Dentist at Ministry of Health B.D.S (2013), Diploma (2016); Nadia M Farrag, Study Director — Professor of Pediatric Dentistry Faculty of Dentistry, Mansoura University; Ahmed H Wahba, Study Director — Lecturer of Pediatric Dentistry Faculty of Dentistry Mansoura University
Locations (1):
- Faculty of Dentistry, Al Mansurah, Egypt

REFERENCES:
- [Background] Leff DR, Nortley M, Dang V, Bhutiani RP. The effect of local cooling on pain perception during infiltration of local anaesthetic agents, a prospective randomised controlled trial. Anaesthesia. 2007 Jul;62(7):677-82. doi: 10.1111/j.1365-2044.2007.05056.x. PMID 17567343
- [Background] Roeber B, Wallace DP, Rothe V, Salama F, Allen KD. Evaluation of the effects of the VibraJect attachment on pain in children receiving local anesthesia. Pediatr Dent. 2011 Jan-Feb;33(1):46-50. PMID 21406147
- [Background] Ram D, Hermida LB, Peretz B. A comparison of warmed and room-temperature anesthetic for local anesthesia in children. Pediatr Dent. 2002 Jul-Aug;24(4):333-6. PMID 12212876
- [Background] Aravena PC, Barrientos C, Troncoso C, Coronado C, Sotelo-Hitschfeld P. Effect of warming anesthetic on pain perception during dental injection: a split-mouth randomized clinical trial. Local Reg Anesth. 2018 Feb 22;11:9-13. doi: 10.2147/LRA.S147288. eCollection 2018. PMID 29503582